CLINICAL TRIAL: NCT03367364
Title: Patient Education Bundle vs. Nurses Feedback and Coaching to Prevent Missed Doses of Venous Thromboembolism (VTE) Prophylaxis: A Crossover, Cluster Randomized Controlled Trial
Brief Title: Patient Education Bundle vs. Nurses Feedback and Coaching to Prevent Missed Doses of VTE Prophylaxis
Acronym: ENACT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: IRB00157201; DI-1603-34596 (Other Grant/Funding Number: PCORI)
Record Dates: First submitted 2017-12-05; First posted 2017-12-08 (Actual); Last update posted 2023-03-02 (Actual); Status verified 2021-12

CONDITIONS: Venous Thrombosis (Disorder)
Keywords: Venous Thromboembolism, Deep Venous Thrombosis, Clots
MeSH Terms: conditions — Venous Thrombosis; Venous Thromboembolism | interventions — BEP protocol

STUDY DESIGN:
Intervention Model Description: In the PEB arm, the intervention will include:
  A charge nurse will intervene in real-time via an EHR-triggered alert when there is documentation that a dose of VTE prophylaxis medication is not given for any reason. The charge nurse will speak to the bedside nurse and one of them will provide the patient with the education bundle including one-on-one personalized discussion, supplemented by a 2-page paper handout and patient education video.
  In the NFC arm, the intervention will include:
  Nurse leadership (i.e. managers, directors) will provide data to all nurses on their personal clinical effectiveness with the proportion of doses of VTE prophylaxis administered. The data will have comparisons to their nurse peers on the same floor. Coaching for nurses will include one-on-one conversations with bedside nurses with lower performance than their peers.
Who Masked: Participant, Outcomes Assessor
Masking Description: Within strata, a coin toss (ERH) will be used to randomize floors into either the Patient education bundle arm or the Nurse feedback arm. The VTE prophylaxis medication non-administration dataset provided to the biostatistical team (i.e. outcomes assessors) for analysis will be blinded by treatment arm and department.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patient education bundle (PEB) (Active Comparator): A charge nurse will intervene in real-time via an EHR-triggered alert when there is documentation that a dose of VTE prophylaxis medication is not given for any reason. The charge nurse will speak to the bedside nurse and one of them will provide the patient with the education bundle including one-on-one personalized discussion, supplemented by a 2-page paper handout and patient education video.
  Interventions: Behavioral: Patient education bundle (PEB),
- Nurse feedback and coaching (NFC) (Placebo Comparator): Nurse leadership (i.e. managers, directors) will provide data to all nurses on their personal clinical effectiveness with the proportion of doses of VTE prophylaxis administered. The data will have comparisons to their nurse peers on the same floor. Coaching for nurses will include one-on-one conversations with bedside nurses with lower performance than their peers.
  Interventions: Behavioral: Nurse feedback and coaching (NFC)

INTERVENTIONS:
Behavioral: Patient education bundle (PEB), — A charge nurse will intervene in real-time via an EHR-triggered alert when there is documentation that a dose of VTE prophylaxis medication is not given for any reason. The charge nurse will speak to the bedside nurse and one of them will provide the patient with the education bundle including one-on-one personalized discussion, supplemented by a 2-page paper handout and patient education video.
  Arms: Patient education bundle (PEB)
Behavioral: Nurse feedback and coaching (NFC) — Nurse leadership (i.e. managers, directors) will provide data to all nurses on their personal clinical effectiveness with the proportion of doses of VTE prophylaxis administered. The data will have comparisons to their nurse peers on the same floor. Coaching for nurses will include one-on-one conversations with bedside nurses with lower performance than their peers.
  Arms: Nurse feedback and coaching (NFC)

SUMMARY:
VTE associated harm is underappreciated among hospitalized patients and may be associated with missed doses of VTE prophylaxis medications. In order to ensure best practices, and administer a defect-free VTE prevention nurses must understand and educate patients on the importance of the VTE prophylaxis. We propose to conduct a randomized trial comparing the effect of a validated, real-time patient education bundle (PEB), to a program of nurse feedback and coaching (NFC) provided by nurse leaders.

DETAILED DESCRIPTION:
Missed doses of prescribed Venous Thromboembolism (VTE) pharmacologic prophylaxis is a significant problem. Data on patients admitted to The Johns Hopkins Hospital found approximately 12% of prescribed doses of pharmacologic VTE prophylaxis were not administered. There were several reasons for these missed doses. The leading reason (nearly 60% of missed doses) was patient or family member refusal for any reason.

Based on data collected by the Maryland Health Services Cost Review Commission (HSCRC) in the Maryland hospital-acquired conditions (MHAC) program, during 2011 half of patients who developed confirmed VTE at The Johns Hopkins Hospital were not administered one or more doses of prescribed VTE prophylaxis. These data indicate that missed or refused doses of VTE prophylaxis represent a significant and under-recognized contributor to sub-optimal VTE prophylaxis that will erode the beneficial impact of current efforts to improve rates of VTE prophylaxis ordering by physicians.

As part of a Patient-Centered Outcomes Research Institute (PCORI)-funded project, the investigators have developed a registry of missed doses of VTE prophylaxis that includes data on missed doses of VTE prophylaxis.

Primary hypothesis Both interventions (PEB and NFC) will improve medication administration (as measured by missed doses)

Secondary hypotheses

1. Combining both interventions (PEB and NFC) will decrease patient refusal of VTE prophylaxis
2. Combining both interventions (PEB and NFC) will decrease missed doses for reasons other than patient refusal
3. Overall, PEB intervention will be more effective than NFC in reducing missed doses for any reason:

   1. The PEB intervention will be more effective than NFC in reducing in reducing patient refusal
   2. The NFC intervention will be more effective than PEB in reducing missed doses for other reasons of missed doses other than patient refusal
4. There will be a differential effect on medicine and surgery floors
5. There will be a differential effect by patient level characteristics (race, age, sex)
6. There will be a differential effect on high vs. low performing floors
7. There will be a differential effect dependent on pharmacological dosing regimen (i.e. medication, frequency)
8. There will be an overall decline in the incidence of VTE events (all, DVT, PE)

Design A single institution, crossover, cluster randomized controlled trial (x-cRCT).

Intervention

In the PEB arm, the intervention will include:

A charge nurse will intervene in real-time via an EHR-triggered alert when there is documentation that a dose of VTE prophylaxis medication is not given for any reason. The charge nurse will speak to the bedside nurse and one of them will provide the patient with the education bundle including one-on-one personalized discussion, supplemented by a 2-page paper handout and patient education video.

In the NFC arm, the intervention will include:

Nurse leadership (i.e. managers, directors) will provide data to all nurses on their personal clinical effectiveness with the proportion of doses of VTE prophylaxis administered. The data will have comparisons to their nurse peers on the same floor. Coaching for nurses will include one-on-one conversations with bedside nurses with lower performance than their peers.

ELIGIBILITY:
1. Eligible floors are defined as:

   A. All medical and surgical floors (non- intensive care units) B. 16 total floors (10 medicine, 6 surgery)
2. Eligible Patients are defined as: All patients on assigned floors except:

A. Patient data for those transferred between floors will be excluded. B. Patient data for those on floors during the cross-over time will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9657 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-11-01 (Actual); Study Completion 2018-11-01 (Actual)

PRIMARY OUTCOMES:
Missed doses of VTE prophylaxis | 1 year
  Proportion of VTE prophylaxis doses not administered

SECONDARY OUTCOMES:
Patient refused doses of VTE prophylaxis | 1 year
  Proportion of VTE prophylaxis doses not administered due to patient/family refusal
Missed doses of VTE prophylaxis for reasons other than patient refusal | 1 year
  Proportion of VTE prophylaxis doses not administered due to reasons other than patient/family refusal
VTE events (all VTE, DVT, PE) | 1 year
  Proportion of VTE events recorded
Patient satisfaction | 1 year
  surveys and HCAHPS scores
Nurse Satisfaction | 1 year
  surveys

CONTACTS AND LOCATIONS:
Overall Officials: Elliott R Haut, MD. PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Medical Institutions, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lau BD, Shaffer DL, Hobson DB, Yenokyan G, Wang J, Sugar EA, Canner JK, Bongiovanni D, Kraus PS, Popoola VO, Shihab HM, Farrow NE, Aboagye JK, Pronovost PJ, Streiff MB, Haut ER. Effectiveness of two distinct web-based education tools for bedside nurses on medication administration practice for venous thromboembolism prevention: A randomized clinical trial. PLoS One. 2017 Aug 16;12(8):e0181664. doi: 10.1371/journal.pone.0181664. eCollection 2017. PMID 28813425
- [Background] Lau BD, Streiff MB, Kraus PS, Hobson DB, Shaffer DL, Aboagye JK, Pronovost PJ, Haut ER. Missed Doses of Venous Thromboembolism (VTE) Prophylaxis at Community Hospitals: Cause for Alarm. J Gen Intern Med. 2018 Jan;33(1):19-20. doi: 10.1007/s11606-017-4203-y. No abstract available. PMID 29043537
- [Background] Streiff MB, Carolan HT, Hobson DB, Kraus PS, Holzmueller CG, Demski R, Lau BD, Biscup-Horn P, Pronovost PJ, Haut ER. Lessons from the Johns Hopkins Multi-Disciplinary Venous Thromboembolism (VTE) Prevention Collaborative. BMJ. 2012 Jun 19;344:e3935. doi: 10.1136/bmj.e3935. PMID 22718994
- [Background] Shermock KM, Lau BD, Haut ER, Hobson DB, Ganetsky VS, Kraus PS, Efird LE, Lehmann CU, Pinto BL, Ross PA, Streiff MB. Patterns of non-administration of ordered doses of venous thromboembolism prophylaxis: implications for novel intervention strategies. PLoS One. 2013 Jun 14;8(6):e66311. doi: 10.1371/journal.pone.0066311. Print 2013. PMID 23799091
- [Background] Haut ER, Lau BD, Kraus PS, Hobson DB, Maheshwari B, Pronovost PJ, Streiff MB. Preventability of Hospital-Acquired Venous Thromboembolism. JAMA Surg. 2015 Sep;150(9):912-5. doi: 10.1001/jamasurg.2015.1340. No abstract available. PMID 26222738
- [Background] Streiff MB, Lau BD, Hobson DB, Kraus PS, Shermock KM, Shaffer DL, Popoola VO, Aboagye JK, Farrow NA, Horn PJ, Shihab HM, Pronovost PJ, Haut ER. The Johns Hopkins Venous Thromboembolism Collaborative: Multidisciplinary team approach to achieve perfect prophylaxis. J Hosp Med. 2016 Dec;11 Suppl 2:S8-S14. doi: 10.1002/jhm.2657. PMID 27925423
- [Derived] Haut ER, Owodunni OP, Wang J, Shaffer DL, Hobson DB, Yenokyan G, Kraus PS, Farrow NE, Canner JK, Florecki KL, Webster KLW, Holzmueller CG, Aboagye JK, Popoola VO, Kia MV, Pronovost PJ, Streiff MB, Lau BD. Alert-Triggered Patient Education Versus Nurse Feedback for Nonadministered Venous Thromboembolism Prophylaxis Doses: A Cluster-Randomized Controlled Trial. J Am Heart Assoc. 2022 Sep 20;11(18):e027119. doi: 10.1161/JAHA.122.027119. Epub 2022 Sep 1. PMID 36047732

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-12-15): https://cdn.clinicaltrials.gov/large-docs/64/NCT03367364/Prot_SAP_000.pdf